CLINICAL TRIAL: NCT07055789
Title: Is a Combined Respiratory Muscle Training Intervention, Incorporating Inspiratory and Expiratory Muscle Training, Feasible in Adult Critical Care Patients? A Single Arm Feasibility Trial.
Brief Title: Is Combined Respiratory Muscle Training, Incorporating Inspiratory and Expiratory Training, Feasible in Adult Critical-care Patients?
Status: Suspended | Phase: Not Applicable | Type: Interventional
Why Stopped: Recruitment suspended pending the finalisation of sponsorship documentation.
Sponsor: Royal College of Surgeons, Ireland (Other)
Collaborators: Tallaght University Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 4331
Record Dates: First submitted 2025-05-08; First posted 2025-07-09 (Actual); Last update posted 2025-07-09 (Actual); Status verified 2025-05

CONDITIONS: Critical Illness Myopathy; Critical Illness
Keywords: inspiratory muscle training; expiratory muscle strength training; respiratory muscle training
MeSH Terms: conditions — Critical Illness

STUDY DESIGN:
Intervention Model Description: Single arm feasibility design
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Single arm feasibility of combined respiratory muscle training (Experimental): The participants will undergo a combined respiratory muscle training intervention including both inspiratory and expiratory muscle training.
  Interventions: Other: Combined respiratory muscle training, incorporating both inspiratory and expiratory muscle training

INTERVENTIONS:
Other: Combined respiratory muscle training, incorporating both inspiratory and expiratory muscle training — IMT: Inspiratory Muscle Training EMST: Expiratory Muscle Strength Training RMST: Respiratory Muscle Strength Training In this trial we are combining both IMT and EMST in the intervention group.
  Other Names: IMT; EMST; RMST

SUMMARY:
Background: Respiratory muscle weakness is a recognised consequence of mechanical ventilation in critical care. This weakness can have implications for patients, leading to prolonged mechanical ventilation (MV) and intensive care unit (ICU) length of stay (LOS), with worse mortality and morbidity outcomes. The aim of this trial is to assess the safety and feasibility of a combined respiratory muscle training (RMST) intervention for respiratory muscle strengthening, in adult critical care patients receiving or recently liberated from mechanical ventilation.

Methods: This prospective single-arm feasibility study will be conducted in Tallaght University Hospital (TUH) ICU. Ethical approval will be sought from TUH ethics committee with sponsorship from (RCSI) Royal College of Surgeons Ireland. Informed consent will be sought from all eligible patients. Participants will receive a combined RMST intervention in addition to usual care. The primary feasibility outcomes of recruitment, adherence and retention will be reported. Secondary clinical outcomes of respiratory muscle strength (maximal inspiratory / expiratory pressure) and cough strength (peak cough flow) will be assessed at recruitment and weekly up to week three. Therapist perception of service usability will be assessed using the service usability survey.

ELIGIBILITY:
Inclusion Criteria:

* Patients ≥18years,
* mechanically ventilated for ≥ 24 hours,
* able to initiate spontaneous breaths on MV,
* on suitable levels of respiratory support with ≤.6 FiO2, ≤10 PEEP,
* deemed eligible for MV weaning by ICU consultant or recently extubated (<48 hours),
* alert and collaborative (RASS -2 to +2).

Exclusion Criteria:

* patients deemed medically unfit by the ICU physicians
* pregnant patients or breast feeding patients
* patients with specific pathologies that may impair respiratory muscle function and response to interventions independent of mechanical ventilation and critical care stay
* Patient who have undergone surgical intervention / repair of the diaphragm within 6 months of the trial, diaphragm / hemi-diaphragm paralysis,
* patients unable to consent / collaborate in treatment,
* patients may also be excluded if the ICU physician deems the short disconnection period from MV is unsuitable,
* patients for palliative management or unlikely to survive their critical care episode.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 25 (Estimated)
Dates: Start 2024-10-01 (Actual); Primary Completion 2026-06 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Recruitment Rate Retention and Adherence Rates | Up to 2 years
  The primary outcome measure for this trial are feasibility outcomes:
  Recruitment rate will be calculated by dividing the number recruited by total number of eligible patients identified and multiplying by 100.
Retention Rates | Up to 2 years
  Retention rate will be described as the percentage of patients with follow up data available
Adherence Rates | Up to 2 years
  Adherence rate will be measured as the number of total treatment sessions divided by the number of potential total sessions, multiplied by 100.

SECONDARY OUTCOMES:
Service Usability Scale. | Up to 2 years
  Staff acceptability of delivering the intervention will assessed using the service usability scale. The scale assess's ten domains of service usability with a score of 1 to 5 denoting strong disagreement (1) up to strong agreement (5)
Inspiratory Muscle Strength | Up to 2 years
  Inspiratory muscle strength will be assessed using Maximal Inspiratory Pressure (MIP): Clinical variability in maximal inspiratory pressure in response to intervention. This will be measured in cmH2O
Expiratory Muscle Strength | Up to 2 years
  Expiratory muscle strength will be assessed using Maximal Expiratory Pressure (MEP). Clinical variability in clinical markers of maximal expiratory pressure in response to intervention. This will be measured in cmH2O
Cough strength | Up to 2 years
  Peak Cough Flow (PCF) will be used to assess cough strength: Clinical variability in peak cough flow will be measured in response to intervention. This measurement unit is L/min.

CONTACTS AND LOCATIONS:
Overall Officials: Eimear McCormack, Principal Investigator — Tallaght University Hospital & Royal College of Surgeons Ireland; Yvelynne Kelly, Doctor, Principal Investigator — Tallaght University Hospital
Locations (1):
- Tallaght University Hospital, Dublin, Tallaght, Ireland

IPD SHARING:
Plan to Share IPD: No